CLINICAL TRIAL: NCT01486823
Title: An Open-label, Single-dose Bioavailability Study of MLDL1278A After Subcutaneous and Intravenous Administration in Healthy Subjects
Brief Title: Bioavailability Study of MLDL1278A After Subcutaneous and Intravenous Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 11-BI-204-02
Record Dates: First submitted 2011-11-22; First posted 2011-12-07 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
MeSH Terms: interventions — MLDL1278A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (Experimental)
  Interventions: Drug: MLDL1278A
- Cohort B (Experimental)
  Interventions: Drug: MLDL1278A

INTERVENTIONS:
Drug: MLDL1278A — Single intravenous dose of 360 mg MLDL1278A followed by a single subcutaneous dose of 360 mg MLDL1278A.
  Arms: Cohort A
Drug: MLDL1278A — Single subcutaneous dose of 360 mg MLDL1278A.
  Arms: Cohort B

SUMMARY:
This is a study in healthy volunteers designed to investigate the PK following intravenous and subcutaneous administration of MLDL1278A (also known as BI-204). The bioavalialbility of MLDL1278A after subcutaneous administration will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Adult males/females aged 18 to 55 years inclusive at screening;
* Subjects who are between 18.0 and 30.0 kg/m2 body mass index (BMI) inclusive and weigh between 55.0 and 100.0 kg inclusive;

Exclusion Criteria:

* Any clinically relevant disease or disorder (past or present), which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study;
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, coagulation, urinalysis, vital signs or ECG at baseline, which, in the opinion of the investigator, may put the subject at risk because of his participation in the study;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of MLDL1278A. | Up to 70 days post administration.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of MLDL1278A. | Up to 70 days post administration.
Plasma clearance (CL) of MLDL1278A. | Up to 70 days post administration.
Number of participants with an anti therapeutic antibody (ATA) response. | Up to 140 days post administration.
Number of participants with adverse events. | Up to 140 days post administration.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom